CLINICAL TRIAL: NCT06098599
Title: A Multicenter, Randomized, Open-lable, Single-dose, Two-cycle, Double-cross Bioequivalence Study Comparing the Pharmacokinetic Profile of LY01612 and CAELYX® in Chinese Subjects With Advanced Breast Cancer
Brief Title: Comparing the Pharmacokinetic Profile of LY01612 and CAELYX® in Chinese Subjects With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY01612/CT-CHN-102
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxorubicin hydrochloride liposome injection(LY01612) (Experimental): 20mg/10mL, 50mg/m2, intravenously for 90min (±3min) with an infusion pump on day 1 and day 29 of the trial.
  Interventions: Drug: Doxorubicin hydrochloride liposome injection
- Doxorubicin hydrochloride liposome injection(CAELYX®) (Active Comparator): 20mg/10mL, 50mg/m2, intravenously for 90min (±3min) with an infusion pump on day 1 and day 29 of the trial
  Interventions: Drug: Doxorubicin hydrochloride liposome injection

INTERVENTIONS:
Drug: Doxorubicin hydrochloride liposome injection — Doxorubicin hydrochloride liposome injection was administered intravenously for 90min (±3min) with an infusion pump on day 1 and day 29 of the trial. Doxorubicin hydrochloride liposome injection was diluted with 250mL 5% glucose injection.

SUMMARY:
A multicenter, randomized, open-lable, single-dose, two-cycle, double-cross bioequivalence study comparing the pharmacokinetic profile of LY01612 (Doxorubicin hydrochloride liposome injection) and CAELYX® in Chinese subjects with advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent;
2. Patients aged ≥18 years and ≤75 years with locally advanced or metastatic breast cancer diagnosed by histology or cytology，and who may benefit from monotherapy of Doxorubicin liposomes;
3. Life expectancy of at least 3 months; Eastern Cooperative Oncology Group (ECOG) performance status (PS)<2;
4. adequate bone marrow function [leukocyte ≥3,000/mm3, absolute neutrophil count (ANC) ≥1,500/mm3, hemoglobin ≥90g/L, and platelet count ≥90,000/mm3；
5. adequate renal function (serum creatinine ≤1.5×Institutional upper limit of normal (ULN));
6. adequate coagulation function [prothrombin time (PT), activated partial thromboplastin time (APTT) ≤1.5×ULN];
7. adequate hepatic function [aspartate aminotransferase (AST), alanine aminotransferase (ALT) level ≤ 2.5×ULN (or ≤5×ULN for subjects with liver metastases), and total bilirubin level ≤ 1.5×ULN (or ≤ 3×ULN for subjects with liver metastases).

Exclusion Criteria:

1. Patients with a diagnosis of severe cardiovascular, lung, liver, kidney, gastrointestinal, endocrine, immune system, skin, musculoskeletal, neurological or psychiatric conditions that the researchers did not consider appropriate for inclusion;
2. With a history of myocardial infarction, unstable angina pectoris, coronary revascularization, New York Heart Association (NYHA) grade ≥Ⅱ cardiac insufficiency, severe pericardial disease, and severe unstable ventricular arrhythmia, cerebrovascular accident or transient cerebral ischemia or pulmonary embolism within 6 months before randomization;
3. Unstable brain metastases;
4. Electrocardiogram (ECG) QTC >480ms; left ventricular ejection fraction <50% or below the lower limit of study center value;
5. The total cumulative dose of doxorubicin was ﹥350mg/m2 before screening；
6. Persistent or active infection requiring systemic treatment;
7. Pregnancy or breast feeding;
8. Other situations that investigators consider as contra-indication for this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
plasma maximum concentration (Cmax) of encapsulated doxorubicin. | from baseline to day 56
Area under Plasma d concentration-time curves of encapsulated doxorubicin | from baseline to day 56
plasma maximum concentration (Cmax) of unencapsulated doxorubicin. | from baseline to day 56
Area under Plasma concentration-time curves of unencapsulated doxorubicin. | from baseline to day 56

SECONDARY OUTCOMES:
plasma maximum concentration（Cmax） of total doxorubicin； | from baseline to day 56
Area under plasma concentration-time curves of total doxorubicin； | from baseline to day 56
Partial area under plasma concentration-time curves （AUC0-48h and AUC48h-t）of encapsulated doxorubicin | from baseline to day 56
Encapsulated doxorubicin、unencapsulated doxorubicin and total doxorubicin Tmax | from baseline to day 56
Encapsulated doxorubicin、unencapsulated doxorubicin and total doxorubicin t1/2z | from baseline to day 56
Adverse event | from baseline to day 56

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: No